CLINICAL TRIAL: NCT05273775
Title: A Single-center, Single-arm, Open-label, Fixed-sequence, Self-controlled Study of the Effects of HRS5091 on the Pharmacokinetics of Midazolam, S-warfarin, Omeprazole, Digoxin and Rosuvastatin in Healthy Volunteers
Brief Title: A Pharmacokinetic Study to Evaluate the Drug Interaction Between HRS5091 and Probe Drugs in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HRS5091-102
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Midazolam; Warfarin; Vitamin K 1; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Single-center, single arm, open-label, fixed sequence, self-control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): HRS5091 + probe drugs (Midazolam Maleate Tablets+Warfarin Sodium Tablets+ Omeprazole Enteric Capsules+ Digoxin Tablets+ Rosuvastatin Calcium) + Vitamin K1 Tablets
  Interventions: Drug: HRS5091 Tablets; Drug: Midazolam Maleate Tablets; Drug: Warfarin Sodium Tablets; Drug: Omeprazole Enteric Capsules; Drug: Vitamin K1 Tablets; Drug: Digoxin Tablets; Drug: Rosuvastatin Calcium Tablets

INTERVENTIONS:
Drug: HRS5091 Tablets — HRS5091 Tablets once daily
Drug: Midazolam Maleate Tablets — Midazolam Maleate Tablets single dose
Drug: Warfarin Sodium Tablets — Warfarin Sodium Tablets single dose
Drug: Omeprazole Enteric Capsules — Omeprazole Enteric Capsules single dose
Drug: Vitamin K1 Tablets — Vitamin K1 Tablets once daily
Drug: Digoxin Tablets — Digoxin Tablets single dose
Drug: Rosuvastatin Calcium Tablets — Rosuvastatin Calcium Tablets single dose

SUMMARY:
This is a drug-drug interaction study conducted in healthy volunteers to evaluate the effect of HRS5091 on CYP3A4, CYP2C9, CYP2C19, P-gp, BCRP and OATP1B1, using midazolam, s-warfarin, omeprazole, digoxin and rosuvastatin as probe drugs.

ELIGIBILITY:
Inclusion Criteria:

1. The subject can communicate well with the researcher, understand and comply with the requirements of this study, and understand and sign the informed consent;
2. Healthy subjects aged 18~50 (including 18 and 50 years old);
3. Body weight ≥ 50 kg, body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26 kg/m2) (BMI= weight (kg)/height2 (m2));
4. Give informed consent not to have a family plan for six months after the last dose, and agree to take effective contraception.

Exclusion Criteria:

1. Has the medicine or food allergy history, or is the allergic constitution person;
2. Inability to swallow, chronic diarrhea and intestinal obstruction, or the presence of a variety of other factors affecting drug use and absorption;
3. QTCF > 450 ms in 12-lead ECG examination or other abnormal conditions judged by the researchers to have clinical significance;
4. Hepatitis B surface Antigen (HBSAG), Hepatitis C virus antibody, human immunodeficiency virus (HIV) antibody, syphilis antibody test positive;
5. Those who smoked more than 5 cigarettes per day within 3 months before screening and could not stop using any tobacco products during the trial period;
6. Regular drinkers who had consumed more than 14 units of alcohol per week (1 unit = 285 ml of beer, 25 ml of spirits, or 100 ml of wine) during the six months prior to screening and could not stop using any alcoholic product during the trial; positive Breath test for alcohol;
7. Having a history of drug abuse, drug dependence (consultation) or positive urine drug abuse screening before drug administration;
8. Anyone who has undergone any surgery within 6 months prior to screening;
9. Clinical trial participants who have participated in any drug or medical device within 3 months prior to screening (subject to the intervention of the experimental drug or medical device);10.Blood donation (or blood loss) within 3 months before screening and the amount of blood donation (or blood loss)≥400 ml, or receiving blood transfusion.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Cmax，PK parameters of midazolam, s-warfarin, omeprazole, digoxin, rosuvastatin before and after oral administration of HRS5091 | Days 1-27
AUC0-t，PK parameters of midazolam, s-warfarin, omeprazole, digoxin, rosuvastatin before and after oral administration of HRS5091 | Days 1-27
AUC0-∞，PK parameters of midazolam, s-warfarin, omeprazole, digoxin, rosuvastatin before and after oral administration of HRS5091 | Days 1-27

SECONDARY OUTCOMES:
Tmax，PK parameters of midazolam, s-warfarin, omeprazole, digoxin, rosuvastatin before and after oral administration of HRS5091 | Days 1-27
t1/2，PK parameters of midazolam, s-warfarin, omeprazole, digoxin, rosuvastatin before and after oral administration of HRS5091 | Days 1-27
CL/F，PK parameters of midazolam, s-warfarin, omeprazole, digoxin, rosuvastatin before and after oral administration of HRS5091 | Days 1-27
Vz/F，PK parameters of midazolam, s-warfarin, omeprazole, digoxin, rosuvastatin before and after oral administration of HRS5091 | Days 1-27
Number of subjects with adverse events and severity of adverse events | Up to 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided